CLINICAL TRIAL: NCT05078099
Title: Eye-tracking Based Amblyopia Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovaSight (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS-00101-R01
Record Dates: First submitted 2021-09-25; First posted 2021-10-14 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2021-09

CONDITIONS: Amblyopia
Keywords: Amblyopia; Lazy eye; Binocular treatment; Dichoptic treatment; Eye tracking; Visual acuity; Stereoacuity; Adherence
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: Single-arm prospective
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm - Binocular CureSight (Experimental): Using binocular treatment device 90 min a day 5 times a week for 12 weeks following by 90 min a day 3 times a week for additional 12 weeks
  Interventions: Device: CureSight

INTERVENTIONS:
Device: CureSight — Binocular eye-tracking-based passive home treatment system delivering personalized amblyopia therapy

SUMMARY:
An Eye-Tracking-Based Binocular Amblyopia Technology Improves Both Visual Acuity and Binocularity

Screening A child is considered for the study after undergoing a standard of care and study-specific eye examinations (by a study investigator as part of the standard of care) that identify amblyopia appearing to meet the eligibility criteria. The study will be discussed with the child's parent(s) or guardian(s) (referred to subsequently as parent (s)). Parent(s) who express an interest in the study will be given a copy of the informed consent form to read. Written informed consent must be obtained from a parent and child prior to performing any study-specific procedures that are not part of the child's routine care.

On screening visit, eligibility assessment, medical history, Demographic data, Refraction and Cycloplegia, Demonstration suitability using the CureSight, ATS Diplopia Questionnaire, Symptom Survey Distance VA Testing, Ocular Alignment Testing, Near VA Testing, Stereoacuity Testing- Titmus Fly, Eye movement exams (optional), Contrast sensitivity (optional), Reading rest (optional).

All eligible subjects enrolled in the study will be followed for 24 weeks of training followed by 52 weeks of follow-up.

24 weeks: Binocular treatment 90 minutes per day, 5 days per week for 12 weeks followed by 90 minutes per day, 3 days per week for an additional 12 weeks

Follow up visits

* Visit 1: 4 weeks ± 1 week
* Visit 2: 8 weeks ± 1 week
* Visit 3: 12 weeks ± 1 week
* Visit 4: 24 weeks ± 1 week (primary endpoint)
* Optional Visit 5: 52 weeks ± 1 week (exploratory outcome, including retainment of improvement; and additional exploratory outcomes)

DETAILED DESCRIPTION:
The Study Purpose is to evaluate the efficacy and safety of a novel binocular eye-tracking-based passive home treatment system delivering personalized amblyopia therapy.

Methods: Real-time foveal area blur was induced on the dominant eye of 20 participants (aged 4-15 years) with anisometropic, strabismic (<5 PD) or mixed amblyopia. Subjects were trained over 12 weeks with 5 weekly sessions and then for an additional 12 weeks with 3 weekly sessions. Primary outcome was the improvement in best-corrected visual acuity (BCVA) and stereo acuity. Secondary outcomes were adherence, improvement persistence, and patient-reported comfort.

Screening A child is considered for the study after undergoing a standard of care and study-specific eye examinations (by a study investigator as part of the standard of care) that identify amblyopia appearing to meet the eligibility criteria. The study will be discussed with the child's parent(s) or guardian(s) (referred to subsequently as parent (s)). Parent(s) who express an interest in the study will be given a copy of the informed consent form to read. Written informed consent must be obtained from a parent and child prior to performing any study-specific procedures that are not part of the child's routine care.

On screening visit, eligibility assessment, medical history, Demographic data, Refraction and Cycloplegia, Demonstration suitability using the CureSight, ATS Diplopia Questionnaire, Symptom Survey, Distance VA Testing, Ocular Alignment Testing, Near VA Testing, Stereoacuity Testing- Titmus Fly, Eye movement exams (optional), Contrast sensitivity (optional), Reading rest (optional).

All eligible subjects enrolled in the study will be followed for 24 weeks:

Binocular treatment 90 minutes per day, 5 days per week for 12 weeks followed by 90 minutes per day, 3 days per week for an additional 12 weeks

Follow up visits

* Visit 1: 4 weeks ± 1 week
* Visit 2: 8 weeks ± 1 week
* Visit 3: 12 weeks ± 1 week
* Optional Visit 5: 52 weeks ± 1 week (exploratory outcome, including retainment of improvement; and additional exploratory outcomes)
* For each individual subject, clinician's decision regarding: continue treatment by patching or terminate treatment Treatment cessation and follow-up; or, Treatment continuation (patching)
* Visit 4: 24 weeks ± 1 week (primary endpoint)

The call center will be comprised of NovaSight personnel, protected by a firewall. For the patching group subjects, the call center personnel will contact all subjects' guardians at 1 week (3 to 7 days) to encourage initial compliance with treatment.

For the CureSight treatment group, the call center will contact the subjects' guardians in order to:

1. Assist first time setup at home over the phone
2. Provide technical support by phone in case of system malfunction or any other query or problem appearing during treatment
3. Respond to compliance notifications of the software and contact the subject's guardians when needed in order to encourage compliance
4. Answer any questions that arise by the subjects or guardians. Permission for such contacts will be included in the Informed Consent Form. The call center personal will be exposed to the following details, contact information, email and phone number.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met for a child to be enrolled in the study:

1. Age 4 to 40 years male and female
2. Amblyopia associated with strabismus, anisometropia, or both (previously treated or untreated)
3. Must have refractive error correction (based on a cycloplegic refraction completed within the last 7 months)
4. Spectacle correction meeting the above criteria must be worn For at least 16 weeks OR until distance VA stability is documented (defined as <0.1 logMAR change by the same testing method measured on 2 consecutive exams at least 8 weeks apart).
5. VA, measured in each eye without cycloplegia in current spectacle correction using the Lea symbol per ATS VA protocol for children < 7 years and the EETDRS VA protocol for children ≥ 7 years on a study-approved device displaying single surrounded optotypes, as follows:

   1. Visual acuity in the amblyopic eye <1.0 logMAR (20/200)
   2. Best-corrected dominant-eye VA <0.2
   3. Interocular difference ≥ 2 logMAR lines
6. Heterotropia with a near deviation of <5∆ (measured by SPCT) in habitual correction (Angles of ocular deviation >4∆ are not allowed because large magnitudes of the deviation would compromise successful alignment of the dichoptic stimuli.)
7. Passing a dedicated 10 min in-clinic performance ability test to assure suitable eye tracking performance (validity of eye tracking data >90% and successful calibration process).

7. Subjects and families eligible for clinic visits over duration of study.

8. Subject in general good health and able, as per investigator decision, to comply with study visits and protocol procedures and wear refractive correction and has access to wireless internet at home which is able to support the CureSight treatment (loaned by sponsor).

9. Signed and dated informed consent form.

10. Parent and participant understand and are willing to comply with study procedures and will be available for the duration of the study.

Exclusion Criteria:

1. Myopia greater than -6.00 D. spherical equivalent in either eye.
2. Known skin reactions to patch or bandage adhesives.
3. Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator).
4. Any condition that might interfere with eye tracking, such as ptosis
5. Any reported anatomic ocular anomaly (e.g., small lens opacity, myelinated nerve fiber layer).
6. Previous intraocular or refractive surgery.
7. Heterophoria with a total near deviation of ≥10Δ (measured by PACT

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity of Amblyopic Eye | 24 weeks
  Mean visual acuity change from baseline Using LogMAR LEA symbols optotype for participants < 7 years of age and LEA numbers optotype for participants ≥ 7 years of age
Best-Corrected Visual Acuity of Fellow Eye | 24 weeks
  Mean visual acuity change from baseline Using LogMAR LEA symbols for participants < 7 years of age and LEA numbers for participants ≥ 7 years of age

SECONDARY OUTCOMES:
Adherence | 4, 8, 12, and 24 weeks
  Duration spent using the device divided by the duration of treatment prescribed
Stereoacuity | 4, 8, 12, and 24 weeks
  Mean stereoacuity change from baseline using the Titmus stereo acuity chart
Amblyopic eye best-corrected visual acuity | 4, 8, 12, and 24 weeks
  Mean visual acuity change from baseline Using LogMAR LEA symbols for participants < 7 years of age and LEA numbers for participants ≥ 7 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Wygnanski-Jaffe, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Select A State, Israel

IPD SHARING:
Plan to Share IPD: No
All data requests should be submitted to the corresponding author for consideration.
  Access to de-identified participant data may be made available with publication for non commercial research with a signed data access agreement

REFERENCES:
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=eye-tracking-based-binocular-amblyopia-treatment-improving-both-visual-acuity-and-binocularity-one-year-follow-up&btnG=